CLINICAL TRIAL: NCT05482620
Title: Parallel-group, Randomized Controlled Trial to Test the Effectiveness of a Nordic Walking Program in Patients With Asthma
Brief Title: Effectiveness of a Nordic Walking in Patients With Asthma.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade da Coruña (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (SEPAR), Spain (Unknown); Colexio Oficial de Fisioterapeutas de Galicia (COFIGA), Spain (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NORWALKAS RCT
Record Dates: First submitted 2022-06-29; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2021-10

CONDITIONS: Asthma
Keywords: Asthma; Physical Therapy, Modalities; Physical Therapy, Speciality; Nordic Walking; Patient Education as Topic; Walk Test; Randomized Controlled Trial
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only investigator making evaluation is blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group (Experimental): Study group following Nordic walking program and educational sessions and usual care (medical visits, medication, etc).
  Interventions: Procedure: Nordic walking program; Procedure: Educational sessions and usual care
- Control Group (Active Comparator): Group that will only receive educational sessions and usual care (medical visits, medication, etc).
  Interventions: Procedure: Educational sessions and usual care

INTERVENTIONS:
Procedure: Nordic walking program — Nordic walking program will consist of three training sessions per week, during eight weeks. Each session will last approximately 60 minutes, including warm-up, the intervention itself and cool-down. Intervention will consist in a 30 minutes Nordic walking, working at 70-85% of maximal heart rate, measured with a Polar pulsometer. Intervention will be delivered in groups (six patients per group as maximum), in designed circuits placed in A Coruña city.
  Arms: Study Group
Procedure: Educational sessions and usual care — Educational sessions will consist in three classes, about 60 minutes each. In these classes, participants will learn about their pulmonary system, asthma disease, asthma diagnosis, asthma classification, asthma exacerbations and triggers, types of medications, how to take inhalers, how to measure PEF (peak expiratory flow), how to control the environment in order to prevent exacerbations, healthy-lifestyle recommendations and the importance of an active lifestyle, what to do in case of asthma emergency, and how to do required data from patients to note in their Patient's Diary (one of the evaluation tools). Usual care implies following the current therapeutic plan and revisions planned by their specialist/GP.

SUMMARY:
A parallel group, randomized controlled trial to compare the effectiveness of an eight-week Nordic walking program plus three educational sessions and usual care in contrast to three educational sessions and usual care in patients with asthma.

The researchers hypothesize that Nordic walking program plus educational sessions and usual care is superior to educational sessions and usual care in terms of exercise tolerance, physical activity, asthma and symptoms control, dyspnea, lung function, handgrip strength, quality of life, quality of sleep, rate of medication intake, treatment adherence, and healthcare use in patients with asthma

DETAILED DESCRIPTION:
Sample size was calculated considering a minimum clinically important difference (MCID) of 26 meters and a standard deviation of 45.49 meters. With a power of 80%, an alpha level of 0.05 and supposing a dropout rate of 15%, a total of 114 patients, 57 in each group, are required.

Patients will be recruited from Pulmonology and Allergology services of University Hospital Complex of A Coruña, Pulmonology service of HM Modelo Hospital (A Coruña) and primary care centres in Coruña.

Nordic walking and educational sessions will be conducted in A Coruña city. Exercise tolerance, physical activity, asthma and symptoms control, dyspnea, lung function, handgrip strength, quality of life, quality of sleep, rate of medication intake, treatment adherence, and healthcare use will be measured at baseline, and then at two (post-intervention), three and six months. Respiratory muscle strength will be measure at baseline to characterize the sample. Any adverse effect occurring during evaluation or intervention will be recorded and analysed.

Data distribution will be check with Kolmogorov-Smirnov test. Quantitative data will be expressed as mean and standard deviation when normally distributed and as a median and quartiles (Q1-Q3) when no normally distributed. To compare outcomes between Nordic walking group (NWG) and control group (CG), it will be calculated an ANOVA test for repeated measures or a Kruskal-Wallis test.

Also, qualitative analysis will be made to get information about NWG experience: the way to deal with the disease, satisfaction with the intervention given, perceived progress in management of disease after intervention. Qualitative information will be collected from focus groups. The interview will be recorded, transcript, and re-read by two of the investigators to generate codes and, afterwards, themes. These themes will be named and defined. Absolut and relative frequencies will be analysed from each theme. Inter-rate agreement will be measured through agreement percentages calculated as number of thematic units in which evaluators agree divided by total number of units; and through Kappa of Cohen, considering >0.81 almost a perfect agreement.

ELIGIBILITY:
Inclusion Criteria:

* Being ≥18 years old.
* Present an asthma diagnosis.
* People that desires participate in the study.
* People able to sign the informed consent.

Exclusion Criteria:

* People with other respiratory pathologies.
* Smokers.
* Asthma exacerbation in the last four weeks.
* Heart failure in the last six months.
* Cardiac arrhythmia with IIIb or superior grade in Lown scale.
* Respiratory infection in the last four weeks.
* Gait disorders that impaired the Nordic walking activity.
* Comorbidities that entail reduced exercise capacity: significant anaemia, electrolyte imbalance, or hyperthyroidism.
* People that follow training sessions of more than 30 minutes per day with a moderate or vigorous intensity.
* People that have followed in last three months a pulmonary rehabilitation program.
* Pregnant and lactating women.
* People meeting exclusion criteria to perform cardiovascular exercise following American Heart Association (AHA).
* People meeting exclusion criteria for 6MWT following ATS/ERS criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2022-06-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Six-minute walk test (6MWT) distance | At baseline, and at two (post-intervention), three and six months.
  Change in the 6MWT distance. The 6MWT will be performed according to the American Thoracic Society / European Respiratory Society recommendations (ATS/ERS).

SECONDARY OUTCOMES:
Number of repetitions in the one-minute sit to stand test (1MSTST) | At baseline, and at two (post-intervention), three and six months.
  Change in number of repetitions of 1MSTST.
Number of steps per day | At baseline, and at two (post-intervention), three and six months.
  Change in number of steps per day measured by accelerometry with DynaPort ® MM+.
Average of steps per week | At two months after baseline measures (post-intervention), at three and six months.
  Analysed through "Patient's Diary", in where they must register daily number of steps walked.
Time lying down | At baseline, and at two (post-intervention), three and six months.
  Change in time lying down measured by accelerometry with DynaPort® MM+.
Time sitting | At baseline, and at two (post-intervention), three and six months.
  Change in time sitting measured by accelerometry with DynaPort® MM+.
Time standing up | At baseline, and at two (post-intervention), three and six months.
  Change in time standing up measured by accelerometry with DynaPort® MM+.
Time walking | At baseline, and at two (post-intervention), three and six months.
  Change in time walking measured by accelerometry with DynaPort® MM+.
Kilocalories consumed | At baseline, and at two (post-intervention), three and six months.
  Change in kilocalories consumed measured by accelerometry with DynaPort ® MM+.
Metabolic equivalent of task (MET) consumed | At baseline, and at two (post-intervention), three and six months.
  Change in MET consumed measured by accelerometry with DynaPort ® MM+ and International Physical Acitvity Questionnaire, short form (IPAQ).
Metabolic equivalent of task (MET) consumed | At baseline, and at two (post-intervention), three and six months.
  Change in MET consumed measured by International Physical Acitvity Questionnaire, short form (IPAQ).
Level of physical activity | At baseline, and at two (post-intervention), three and six months.
  Change in category level of physical activity (low (worst level of physical activity), moderate or high) in function of MET-minutes/week, measured by International Physical Activity Questionnaire, a cualitative and quantitative scale.
Asthma-related symptoms and asthma control | At baseline, and at two (post-intervention), three and six months.
  Change in Control of Allergic Rhinitis and Asthma Test (CARAT) results, validated in patients with asthma and in Spanish population. The range of possible scores is 0-30, being 0 the complete absence of control.
Asthma-related symptoms and asthma control | At baseline, and at two (post-intervention), three and six months.
  Change in Test of Adherence to Inhalers (TAI) results, validated in patients with asthma and in Spanish population. Score range is from 10 to 50, being 10 the worst score.
Asthma-related symptoms and asthma control | At two months after baseline measures (post-intervention), at three and six months.
  Analysed through "Patient's Diary", in where they must register some data that the researchers will analyse afterwards (dyspnea measured using Borg's modified scale, in expectoration, cough, feeling of chest wheezing, medicine intake, unscheduled medical consultations, emergency visits, PEF diary measure with a peak flow meter).
Dyspnea | At baseline, and at two (post-intervention), three and six months.
  Change in dyspnea measured with Modified Medical Research Council scale (mMRC). Scores range from 0 to 4, being 0 the best punctuation.
Pulmonary function | At baseline, and at two (post-intervention), three and six months.
  Forced spirometry (Datospir® 120C, Sibelmed, Barcelona, Spain): to analyse changes in forced expiratory volume in first second (FEV1), forced vital capacity (FVC), FEV1/FVC. Following international recommendations of American Thoracic Society / European Respiratory Society (ATS/ERS).
Handgrip Strength | At baseline, and at two (post-intervention), three and six months.
  Change in handgrip strength measured through handgrip dynamometry with Jamar® Hydraulic Hand dynamometer (Performance Health, Warrenville, IL, USA), following the international recommendations (Mathiowetz et al., 1985).
Health Related Quality of Life | At baseline, and at two (post-intervention), three and six months.
  Change in EuroQol 5-dimensions 5-levels (EQ-5D-5L) questionnaire results, validated in people with asthma and in Spanish population. Each dimension can be scored from level 1 (no problems in a specific dimension) to level 5 (extreme problems in a specific dimension).
Health Related Quality of Life | At baseline, and at two (post-intervention), three and six months.
  Changes in mini-Asthma Quality of Life Questionnaire (miniAQLQ) results, validated in Spanish. It is a 15-questions questionnaire, with seven possible responses, ranged in a 7-point scale from 1='extremely bothered' to 7='not bothered at all' . All questions are equally weighted and the overall score is the mean of the 15 responses. So, the final score can range also from 1 to 7, being 1 the worst punctuation.
Qualitative changes in the physical activity done in patient's daily life. | At two months after baseline measures (post-intervention), at three and six months.
  Changes in physical activity registered by patients in their Patient's Diary will be analysed.
Qualitative changes in self-perception of mood in patient's daily life. | At two months after baseline measures (post-intervention), at three and six months.
  Changes in self-perception of mood registered by patients in their Patient's Diary will be analysed.
Quality of sleep | At baseline, and at two (post-intervention), three and six months.
  Change in Pittsburgh Quality Sleep Index (PQSI) results, validated in Spanish population. The PSQI global score has a possible range of 0 to 21 points, being 0 the best score.
Medication adherence and recommendations compliance | At two months after baseline measures (post-intervention), three and six months.
  Adherence will be assessed by analysing different items that the participants should note in their Patients's Diary, in order to determine the treatment and recommendations compliance.

OTHER OUTCOMES:
Medicine intake | At two months after baseline measures (post-intervention), at three and six months.
  Using information noted by patients in their Patient's diary.
Health care use | At two months after baseline measures (post-intervention), at three and six months.
  Information noted by patients in their Patient's diary, relative to unscheduled medical consultations and emergency department visits.
Respiratory Muscle Strength | At baseline
  Maximal inspiratory pressure (PImax) and maximal expiratory pressure (PEmax) will be measured following recommendations of Spanish Society of Pulmonology and Thoracic Surgery (SEPAR) using a digital manometer MicroRPM® (Vyaire Medical GmbH, Hoechberg, Germany), and PUMA® software (Vyaire Medical GmbH, Hoechberg, Germany). No change is expected, so the measure will be only assessed at baseline in order to characterize the sample.
Adverse effects | During intervention, at two months after baseline measures (post-intervention), three and six months.
  Any inconvenience related with intervention, or affecting it, will be registered.
Satisfaction of Nordic walking group with intervention given | At two months after baseline measures (post-intervention).
  It will be assessed with a group interview through focus groups only in Nordic walking intervention group. The interview will be made following a semi structured guide with open-ended questions to try to aboard: the way of affront their disease; experience and satisfaction with the intervention given (facilitators and barriers to their participation) and perceived improvement in asthma management after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Physiotherapy. The University of A Coruña. Campus Universitario de Oza, number 1., A Coruña, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Holland AE, Spruit MA, Troosters T, Puhan MA, Pepin V, Saey D, McCormack MC, Carlin BW, Sciurba FC, Pitta F, Wanger J, MacIntyre N, Kaminsky DA, Culver BH, Revill SM, Hernandes NA, Andrianopoulos V, Camillo CA, Mitchell KE, Lee AL, Hill CJ, Singh SJ. An official European Respiratory Society/American Thoracic Society technical standard: field walking tests in chronic respiratory disease. Eur Respir J. 2014 Dec;44(6):1428-46. doi: 10.1183/09031936.00150314. Epub 2014 Oct 30. PMID 25359355
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151
- [Background] Kendrick KR, Baxi SC, Smith RM. Usefulness of the modified 0-10 Borg scale in assessing the degree of dyspnea in patients with COPD and asthma. J Emerg Nurs. 2000 Jun;26(3):216-22. doi: 10.1016/s0099-1767(00)90093-x. PMID 10839848
- [Background] Fonseca JA, Nogueira-Silva L, Morais-Almeida M, Azevedo L, Sa-Sousa A, Branco-Ferreira M, Fernandes L, Bousquet J. Validation of a questionnaire (CARAT10) to assess rhinitis and asthma in patients with asthma. Allergy. 2010 Aug;65(8):1042-8. doi: 10.1111/j.1398-9995.2009.02310.x. Epub 2010 Feb 1. PMID 20121755
- [Background] Azevedo P, Correia de Sousa J, Bousquet J, Bugalho-Almeida A, Del Giacco SR, Demoly P, Haahtela T, Jacinto T, Garcia-Larsen V, van der Molen T, Morais-Almeida M, Nogueira-Silva L, Pereira AM, Rodriguez MR, Silva BG, Tsiligianni IG, Yaman H, Yawn B, Fonseca JA; WHO Collaborative Center for Asthma and Rhinitis, Montpellier. Control of Allergic Rhinitis and Asthma Test (CARAT): dissemination and applications in primary care. Prim Care Respir J. 2013 Mar;22(1):112-6. doi: 10.4104/pcrj.2013.00012. PMID 23412110
- [Background] Plaza V, Lopez-Vina A, Cosio BG; en representacion del Comite Cientifico del Proyecto TAI. Test of Adherence to Inhalers. Arch Bronconeumol. 2017 Jul;53(7):360-361. doi: 10.1016/j.arbres.2016.08.006. Epub 2016 Oct 15. No abstract available. English, Spanish. PMID 27756657
- [Background] Mathiowetz V, Kashman N, Volland G, Weber K, Dowe M, Rogers S. Grip and pinch strength: normative data for adults. Arch Phys Med Rehabil. 1985 Feb;66(2):69-74. PMID 3970660
- [Background] Hernandez G, Garin O, Dima AL, Pont A, Marti Pastor M, Alonso J, Van Ganse E, Laforest L, de Bruin M, Mayoral K, Serra-Sutton V, Ferrer M; ASTRO-LAB Group. EuroQol (EQ-5D-5L) Validity in Assessing the Quality of Life in Adults With Asthma: Cross-Sectional Study. J Med Internet Res. 2019 Jan 23;21(1):e10178. doi: 10.2196/10178. PMID 30672744
- [Background] Hernandez G, Garin O, Pardo Y, Vilagut G, Pont A, Suarez M, Neira M, Rajmil L, Gorostiza I, Ramallo-Farina Y, Cabases J, Alonso J, Ferrer M. Validity of the EQ-5D-5L and reference norms for the Spanish population. Qual Life Res. 2018 Sep;27(9):2337-2348. doi: 10.1007/s11136-018-1877-5. Epub 2018 May 16. PMID 29767329
- [Background] Juniper EF, Guyatt GH, Cox FM, Ferrie PJ, King DR. Development and validation of the Mini Asthma Quality of Life Questionnaire. Eur Respir J. 1999 Jul;14(1):32-8. doi: 10.1034/j.1399-3003.1999.14a08.x. PMID 10489826
- [Background] Fletcher GF, Ades PA, Kligfield P, Arena R, Balady GJ, Bittner VA, Coke LA, Fleg JL, Forman DE, Gerber TC, Gulati M, Madan K, Rhodes J, Thompson PD, Williams MA; American Heart Association Exercise, Cardiac Rehabilitation, and Prevention Committee of the Council on Clinical Cardiology, Council on Nutrition, Physical Activity and Metabolism, Council on Cardiovascular and Stroke Nursing, and Council on Epidemiology and Prevention. Exercise standards for testing and training: a scientific statement from the American Heart Association. Circulation. 2013 Aug 20;128(8):873-934. doi: 10.1161/CIR.0b013e31829b5b44. Epub 2013 Jul 22. No abstract available. PMID 23877260
- [Background] Van Remoortel H, Raste Y, Louvaris Z, Giavedoni S, Burtin C, Langer D, Wilson F, Rabinovich R, Vogiatzis I, Hopkinson NS, Troosters T; PROactive consortium. Validity of six activity monitors in chronic obstructive pulmonary disease: a comparison with indirect calorimetry. PLoS One. 2012;7(6):e39198. doi: 10.1371/journal.pone.0039198. Epub 2012 Jun 20. PMID 22745715
- [Derived] Vilanova-Pereira M, Jacome C, Rial Prado MJ, Barral-Fernandez M, Blanco Aparicio M, Fontan Garcia-Boente L, Lista-Paz A. Effectiveness of nordic walking in patients with asthma: A study protocol of a randomized controlled trial. PLoS One. 2023 Mar 9;18(3):e0281007. doi: 10.1371/journal.pone.0281007. eCollection 2023. PMID 36893205